CLINICAL TRIAL: NCT02468453
Title: Multi-center, Multi-cohort, Prospective, Open-label Study of VELOS for Treatment of Vascular Skin Disorders
Brief Title: VELOS for the Treatment of Vascular Lesions and Skin Rejuvenation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IH149901
Record Dates: First submitted 2015-05-31; First posted 2015-06-10 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Vascular Lesions; Photoaging
Keywords: velos; Vascular; Rejuvenation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 -facial skin disorders (Experimental): Pulsed dye laser/bipolar radiofrequency (Velos) treatment of facial skin disorders including photo-damage, age spots, lentigos, solar telangiectasia and general facial telangiectasia
  Interventions: Device: velos
- Cohort 2 - leg veins (Experimental): Pulsed dye laser/bipolar radiofrequency (Velos) treatment of leg veins of diameter of at least 1mm, i.e., venulectasia and reticular leg veins.
  Interventions: Device: velos
- Cohort 3-general skin rejuvenation (Experimental): Pulsed dye laser/bipolar radiofrequency (Velos) treatment treatment of general skin rejuvenation including Rosacea, erythematous scars (including acne), and erythematous striae (subjects enrolled in this group must have at least two of the above mentioned treatment indications.
  Interventions: Device: velos
- Cohort 4-improving skin laxity (Experimental): Velos (Bipolar radiofrequency only) treatment for improving skin laxity or skin tightness/firmness
  Interventions: Device: velos

INTERVENTIONS:
Device: velos — VELOS combines 595nm pulsed dye laser energy with bipolar RF energy. The study device can deliver 0.45 to 40 ms laser pulses at a maximum of 25 J/cm2

SUMMARY:
This is a multi-center, multi-cohort, prospective, open-label study of VELOS for treatment of vascular skin disorders. The plan is to enroll up to 60 subjects from up to 3 centers in the US and worldwide. The purpose is to collect data from the use of VELOS.

DETAILED DESCRIPTION:
The primary objective of this trial is to collect data from the use of VELOS in clinical practice under a wide range of treatment parameters variability including RF energy, laser fluence, and laser pulse duration for treating each of the vascular disorders. This will be conducted by documenting the physician selected treatment parameters, as well as the subjects' clinical clearing response, perception of improvement and sensations, through the study treatments and post-treatment(s) follow-up visits.

Optional exploratory objectives: Collection of safety and efficacy data of the Velos with DCD cooling and Velos with contact cooling. The investigator may opt to include in this study noninvasive measurements of erythema, melanin and texture (which may be performed by eg. Chromameter, Mexameter or 3D imaging), and measurements of linear vessel diameters and lesion size.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a healthy Male or Female at least 18 years of age
2. Subject has a vascular (blood vessels) and skin disorders or erythematous scars or erythematous striae or wishes to improve skin laxity or skin firmness. In special cases non-erythematous scars or non-erythematous striae may be allowed as well.
3. Fitzpatrick Skin Type I - VI
4. Subject must be able to read, understand and sign the Informed Consent Form
5. Subject must be willing and able to adhere to the treatment and follow-up schedule and post-treatment care instructions
6. Subject must be willing to have limited sun exposure for the duration of the study, including the follow-up period
7. Subject is willing to have photographs and/or videos taken of the treated area which will be used, de-identified, in evaluations and may be used, de-identified, in presentations and/or publications
8. For female candidates - subject must be post-menopausal, or surgically sterilized, or using a medically acceptable form of birth control during the entire course of the study.

Exclusion Criteria:

1. Subject is pregnant or planning to become pregnant during the study duration. Pregnancy will be assessed by question at screening.
2. Subject has an active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator.
3. Subject has an implant in the treated area (such as metal plates or screws) or an injected chemical substance, including Botox and collagen injections (if the face area is treated).
4. Subject has a known collagen (connective tissue) disorder, vascular disease, scleroderma or other autoimmune disease (i.e. rheumatoid arthritis, lupus).
5. Subject has a history of diseases stimulated by heat or sun exposure, such as recurrent Herpes Simplex in the treated area, unless treatment is conducted following a prophylactic regimen.
6. Subject has a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications.
7. Having or undergoing any form of treatment for active cancer, or having a history of skin cancer or any other cancer in the areas to be treated, including actinic keratosis, presence of malignant or pre-malignant pigmented lesions.
8. Subject is suffering from significant concurrent illness, such as such as cardiac disorders, diabetes (type I or II), or pertinent neurological disorders.
9. Subject has an infection or is suffering from current or has a history of significant skin conditions in the treated area or inflammatory skin conditions, including, but not limited to: photodermatoses, active acne, excessive skin dryness, psoriasis, eczema, rash, rosacea (particularly severe open wound stage), varicella scars, open lacerations or abrasions and active cold sores or herpes sores prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course.
10. Having a known anticoagulative or thromboembolic condition or taking anticoagulation medications one week prior to and during the treatment course (to allow inclusion, temporary cessation of use as per the subject's physician discretion).
11. Use of non-steroidal anti-inflammatory drugs (NSAIDS, e.g., ibuprofen-containing agents) one week before and after each treatment session.
12. Subject has a history of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation.
13. Subject has a history of keloid scarring or of abnormal wound healing.
14. Subject has a known photosensitivity to the study laser wavelength, history of ingesting medications known to induce photosensitivity, or history of seizure disorders due to light.
15. Subject has undergone any surgical, light-based therapy or RF procedures in the treatment area within 3 months of treatment or during the study.
16. Having undergone any other surgery in the treated area within 3 months of treatment (or more if skin has not healed completely) or during the study.
17. Subject has undergone a facial dermabrasion or chemical peel treatment within 3 months of treatment or during the study (if face is treated).
18. Having received Botox/collagen/fat injections or other methods of augmentation with injected or implanted material in the treated area within 9 months of treatment or during the study (if face is treated).
19. Subject has undergone a resurfacing procedure, face lift or eyelid surgery within a year of treatment or during the study (if face is treated).
20. Subject has a tattoo or permanent make-up in the treated area.
21. Subject has systemically used retinoids, antioxidants or medical grade of skin nourishing supplements within 2 months of treatment or during the study.
22. Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
23. Participation in a study of another device or drug within three months prior to enrollment or during the study.
24. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-07-01 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Evidence of leg vein and skin improvement by validated vascular assessment scale and wrinkle assessment scale | up to 3 months after treatment
  Evidence of leg vein and skin improvement by validated vascular assessment scale and wrinkle assessment scale

SECONDARY OUTCOMES:
Number and severity of all complications caused by the laser will be recorded and descriptively tabulated | up to 3 months
Subject Improvement Questionnaire | up to 6 months
Subject assessment of comfort level associated with treatment | day 0, afer 4 weeks, 8 weeks and 12 weeks
  Numerical Response Scale for Rating Pain (NRS)

CONTACTS AND LOCATIONS:
Overall Officials: Shlomit Mann, MSc, Study Director — Syneron Medical
Locations (4):
- United States (4):
  - Scripps Clinic - Carmel Valley, San Diego, California
  - Syneron Candela Institute for Education Clinic, Wayland, Massachusetts
  - Zel Skin & Laser Specialists, Edina, Minnesota
  - Laser and Skin Surgery Center of New York, New York, New York

REFERENCES:
- [Background] Sadick NS, Makino Y. Selective electro-thermolysis in aesthetic medicine: a review. Lasers Surg Med. 2004;34(2):91-7. doi: 10.1002/lsm.20013. PMID 15004818
- [Background] Sadick NS. Combination radiofrequency and light energies: electro-optical synergy technology in esthetic medicine. Dermatol Surg. 2005 Sep;31(9 Pt 2):1211-7; discussion 1217. doi: 10.1111/j.1524-4725.2005.31928. PMID 16176773